CLINICAL TRIAL: NCT02039908
Title: Examining Tolerance to CNS Stimulants in ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MH099030
Record Dates: First submitted 2013-03-07; First posted 2014-01-20 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Tolerance to stimulant medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate 7-day dosing (Active Comparator): During the school year, children in this arm will receive 7-day dosing of medication.
  Interventions: Drug: Methylphenidate
- Methylphenidate 5-day dosing (Active Comparator): During the school year phase, these children will receive 5-day dosing with weekend holidays.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Children will receive a double-blind assessment to determine their optimal starting dose of Concerta. Doses will be adjusted over the course of the school year and inceased if tolerance to the medication is detected.
  Other Names: Concerta

SUMMARY:
Although stimulant medication is a well-established treatment for ADHD, it is often necessary for doctors to increase the dose over time to maintain the benefits of the medication. While medication can be very effective for improving symptoms of ADHD during the first year of use, it has not been found to significantly improve the long term course of children with ADHD. For example, in large research studies, groups of children who take medication for ten years do not have consistently better academic grades than groups of children who never used medication (individual results will vary from child to child).

In order to help children with ADHD achieve the best possible outcomes, it is important for doctors to study why this happens. One possible reason is development of tolerance to the medication. Tolerance means that a drug's effects decrease when it is taken consistently over time, so that an increased dose is needed to continue showing effects. Some doctors believe that children who take stimulant medication for ADHD develop tolerance to it which would explain why benefits may not persist over time, but no research studies have been done to measure whether this occurs. This study aims to see if children show a tolerance effect to stimulant medication and whether that tolerance can be prevented by taking short breaks from the medication called medication holidays.

DETAILED DESCRIPTION:
This is an innovative evaluation of tolerance using an objective measure in an analog classroom. Each subject will complete the a 10-minute math test twice a day for three weeks on optimal dose or placebo, and then be crossed over to the other condition. Within-subject drug/placebo differences will be compared over the three weeks of exposure to assess tolerance in the analog setting.

When school commences, 50% of the sample will be randomized to 7-day-a-week (continuous) dosing and 50% to 5-day-a- week (weekend holidays) dosing to examine the efficacy of prescribed weekend drug holidays for combatting need for dose escalations (tolerance) during the school year.

Participants will be assessed monthly to detect deteriorating functioning. Using a standardized protocol, study physicians will increase dose for subjects in either arm who meet defined impairment thresholds. The difference between the two dosing conditions will inform regarding how best to deal with tolerance in clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of attention-deficit/hyperactivity disorder
* Full Scale IQ above 80

Exclusion Criteria:

* Psychotropic medications for conditions other than ADHD
* Active medical or psychiatric conditions that could be worsened by stimulants
* Diagnosis of Autism or Asperger's Disorder
* Documented intolerance fo methylphenidate or failed trial of OROS MPH

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2013-04; Primary Completion 2018-05 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Pelham, Ph.D., Principal Investigator — Florida International University; James M Swanson, Ph.D., Principal Investigator — Florida International University
Locations (1):
- Florida International University Center for Children and Families, Miami, Florida, United States

REFERENCES:
- [Derived] Pelham WE, Altszuler AR, Merrill BM, Raiker JS, Macphee FL, Ramos M, Gnagy EM, Greiner AR, Coles EK, Connor CM, Lonigan CJ, Burger L, Morrow AS, Zhao X, Swanson JM, Waxmonsky JG, Pelham WE. The effect of stimulant medication on the learning of academic curricula in children with ADHD: A randomized crossover study. J Consult Clin Psychol. 2022 May;90(5):367-380. doi: 10.1037/ccp0000725. PMID 35604744
- See also: Center for Children and Families General Information — http://ccf.fiu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 4 annual cohorts from 2013-2016. Participants could be referred by schools, physicians, or community advertisement; interested parents completed phone screens and a clinic intake to assess inclusionary and exclusionary criteria.
Pre-assignment Details: Because all participants were required to be enrolled in a Summer Treatment Program, some participants withdrew after consenting because they were unable to make the time commitment to the 8-week summer program.
Groups:
- Phase 1-Summer; Medication First, Then Placebo: In the first phase of the study, children participated in a crossover design of placebo and optimal-dose methylphenidate for 13 days in each condition. After a 9-day titration period, the Medication First group received their optimal dose of methylphenidate for 13 days, a 2-day medication/placebo probe, a 2-day washout, then placebo for 13 days and a 2-day medication/placebo probe.
- Phase 1-Summer; Placebo First, Then Medication: In the first phase of the study, children participated in a crossover design of placebo and optimal-dose methylphenidate for 13 days in each condition. After a 9-day titration period, the Placebo First group received placebo for 13 days, a 2-day medication/placebo probe, a 2-day washout, then optimal-dose medication for 13 days and a 2-day medication/placebo probe.
- Phase 2 School Year - 7-Day Dosing: During the school year, all participants took their optimal dose determined in Phase 1 of the study for the entire school year. These partcipants received medication 7-days a week for the entire year.
- Phase 2 School Year; 5-Day Dosing: During the school year, all participants took their optimal dose determined during Phase 1 for the entire school year. These participants received medication on school-days only with drug holidays over weekends.
Period: Phase 1-Summer
Arm/Group | Phase 1-Summer; Medication First, Then Placebo | Phase 1-Summer; Placebo First, Then Medication | Phase 2 School Year - 7-Day Dosing | Phase 2 School Year; 5-Day Dosing
Started | 129 | 138 | 0 | 0
Completed | 116 | 132 | 0 | 0
Not Completed | 13 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 6 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 0 | 0
Period: Phase 2-School Year
Arm/Group | Phase 1-Summer; Medication First, Then Placebo | Phase 1-Summer; Placebo First, Then Medication | Phase 2 School Year - 7-Day Dosing | Phase 2 School Year; 5-Day Dosing
Started (Three participants elected not to continue in the study for the school -year phase.) | 0 | 0 | 121 | 124
Completed | 0 | 0 | 109 | 116
Not Completed | 0 | 0 | 12 | 8
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase 1-Summer: In the first phase of the study, all children participate in a crossover design of placebo and optimal-dose methylphenidate for 13 days in each condition.
Arm/Group | Phase 1-Summer
Number analyzed (Participants) | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 267
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 224
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 237
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 267

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Changes Required Per Protocol
Description: Monthly evaluations of medication efficacy will be used to determine whether dose adjustments are needed due to anticipated tolerance effects.
Time Frame: 10 months
Population: All participants who began Phase 2 were included in analysis
Measure: Mean (Standard Deviation); unit: Number of Increases
Arm/Group | Methylphenidate 7-day Dosing | Methylphenidate 5-day Dosing
Number analyzed (Participants) | 124 | 121
Number of Increases | 1.79 (1.16) | 1.61 (1.08)

2. Secondary Outcome: Time to First Dose Increase
Description: The amount of time elapsed before a child requires a dose increase during the school year will be measured in months.
Time Frame: 10 months
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Methylphenidate 7-day Dosing | Methylphenidate 5-day Dosing
Number analyzed (Participants) | 124 | 121
Months | 3.8 (3.4) | 4.1 (3.5)

3. Secondary Outcome: Endpoint Medication Dose
Description: Dose of medication reported in mg/kg/day
Time Frame: End of Phase 2 School Year
Population: Only participants who completed the entire school year are used in endpoint medication dosing calculations.
Measure: Mean (Standard Deviation); unit: Mg/kg/day
Arm/Group | Methylphenidate 7-day Dosing | Methylphenidate 5-day Dosing
Number analyzed (Participants) | 116 | 109
Mg/kg/day | 1.30 (0.43) | 1.24 (0.41)

ADVERSE EVENTS:
Time Frame: During Phase 1, side effects ratings were collected from parents daily for the first 2 weeks of the summer and weekly for the final 6 weeks of the summer. During Phase 2, side-effects ratings were completed by parents monthly at medication dispensing visits.
Description: Parents completed the Pittsburgh Side Effects Rating Scale, rating each of the most common side effects of stimulant medication on a scale of None, Mild, Moderate, or Severe. Adverse events were counted if parents rated the side effect at the Moderate or Severe level on at least one occasion,
Groups:
- Phase 1-Medication First: In the first phase of the study, children participated in a crossover design of placebo and optimal-dose methylphenidate for 13 days in each condition. After a 9-day titration period, the Medication First group received methylphenidate for 13 days, a 2-day medication/placebo probe, a 2-day washout, then placebo for 13 days and a 2-day medication/placebo probe.
- Phase 1 - Placebo First: In the first phase of the study, children participated in a crossover design of placebo and optimal-dose methylphenidate for 13 days in each condition. After a 9-day titration period, the Placebo First group received placebo for 13 days, a 2-day medication/placebo probe, a 2-day washout, then optimal-dose medication for 13 days and a 2-day medication/placebo probe.
- Phase 2 - 7-Day Dosing: During the school year, all participants took their optimal dose determined in Phase 1 of the study for the entire school year. These participants received medication 7-days a week for the entire year
- Phase 2 - 5-Day Dosing: During the school year, all participants took their optimal dose determined during Phase 1 for the entire school year. These participants received medication on school-days only with drug holidays over weekends.
Arm/Group | Phase 1-Medication First | Phase 1 - Placebo First | Phase 2 - 7-Day Dosing | Phase 2 - 5-Day Dosing
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/138 | 0/121 | 0/124
Serious Adverse Events (participants affected / at risk) | 1/129 | 0/138 | 1/121 | 1/124
Other Adverse Events (participants affected / at risk) | 72/129 | 78/138 | 91/121 | 85/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1-Medication First (N=129) | Phase 1 - Placebo First (N=138) | Phase 2 - 7-Day Dosing (N=121) | Phase 2 - 5-Day Dosing (N=124)
Hospitalized (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Referred by parent for inpatient psychiatric treatment due to comorbid mental health issues.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1-Medication First (N=129) | Phase 1 - Placebo First (N=138) | Phase 2 - 7-Day Dosing (N=121) | Phase 2 - 5-Day Dosing (N=124)
Appetite Loss (Gastrointestinal disorders) | 66 (252) | 72 (265) | 46 (131) | 51 (143) — Moderate or Severe Appetite Loss
Insomnia (General disorders) | 52 (163) | 56 (190) | 46 (118) | 34 (80)
Motor Tics (General disorders) | 17 (23) | 19 (25) | 17 (24) | 14 (19) — Rating of moderate or severe motor tics
Buccal-lingual movements (General disorders) | 15 (27) | 17 (29) | 10 (11) | 16 (20) — Parent rating of moderate or severe buccal-lingual movements
Picking at skin, nailbiting (General disorders) | 37 (83) | 28 (90) | 38 (73) | 37 (91) — Parent rating of moderate or severe picking, nail-biting, etc.
Worried/Anxious (General disorders) | 27 (61) | 30 (66) | 25 (40) | 34 (63) — Parent rating of moderate or severe worry/anxiety
Dull, tired, listless (General disorders) | 27 (56) | 30 (61) | 14 (18) | 19 (32) — Parent rating of moderate or severe dullness/tiredness/listlessness
Headache (General disorders) | 17 (32) | 19 (32) | 15 (24) | 14 (23) — Parent rating of moderate or severe headache
Stomachache (Gastrointestinal disorders) | 23 (51) | 24 (55) | 21 (29) | 17 (25) — Parent rating of moderate or severe stomach ache
Irritability (General disorders) | 42 (97) | 46 (104) | 38 (71) | 36 (62) — Parent rating of moderate or severe irritability
Tearful, depressed (General disorders) | 25 (49) | 27 (53) | 14 (15) | 20 (31) — Parent rating of moderate or severe tearfulness or sadness
Social Withdrawal (General disorders) | 13 (13) | 14 (28) | 5 (6) | 10 (16) — Parent rating of moderate or severe social withdrawal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02039908/Prot_SAP_000.pdf